CLINICAL TRIAL: NCT00638976
Title: INSTANT: INtegrilin Plus STenting to Avoid Myocardial Necrosis Trial
Acronym: INSTANT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Evidence per Attività e Ricerche Cardiovascolari ONLUS (Other)
Responsible Party: Principal Investigator: Dr. Giuseppe Massimo Sangiorgi, PTV Rome
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Fondazione Mediolanum 001/2007
Record Dates: First submitted 2008-03-13; First posted 2008-03-19 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Cardiovascular Disease
Keywords: Eptifibatide; IV eptifibatide; GP IIB/IIIA inhibitors; DES stent
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Eptifibatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.Integrilin, GSK (Other): Pre-procedural use of the Gp IIb/IIIa inhibitor eptifibatide (Integrilin, GSK) vs matched placebo.
  Interventions: Drug: eptifibatide
- 2 (Placebo Comparator): Pre-procedural use of the Gp IIb/IIIa inhibitor eptifibatide (Integrilin, GSK) vs matched placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: eptifibatide — Enrolled patients will be randomized in the catheterization laboratory, after the decision to perform PCI by means of planned implantation of DES >33 mm in length in the same coronary vessel, to IV placebo or IV eptifibatide (double bolus [180 microg/kg] followed by infusion [2 microg/kg per minute] for 18 to 24 hours after the procedure
  Arms: 1.Integrilin, GSK
Drug: placebo — Enrolled patients will be randomized in the catheterization laboratory, after the decision to perform PCI by means of planned implantation of DES >33 mm in length in the same coronary vessel, to IV placebo or IV eptifibatide (double bolus [180 microg/kg] followed by infusion [2 microg/kg per minute] for 18 to 24 hours after the procedure
  Arms: 2

SUMMARY:
Randomized, blind controlled, Multicenter, spontaneous, prospective trial, roughly 20 enrolling centers in Italy, placebo and active drug supply given by GlaxoSmithKline (GSK).

DETAILED DESCRIPTION:
The Objective of the trial is compare the efficacy and, secondarily, the safety and effectiveness of pre-procedural use of the Gp IIb/IIIa inhibitor eptifibatide in comparison to placebo in patients with diffuse CAD undergoing multiple DES implantation.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this study must meet all of the following criteria:

* Male or female able to understand and sign a witnessed informed consent
* Age ≥ 18 yo
* Patients with stable (CCS 1-4) or unstable angina pectoris (but with the most recent anginal episode occurring >48 hours before the procedure) or documented silent ischemia
* Stable Hemodynamic conditions (systolic BP > 100 HR > 40 < 100).
* No clinical and ECG changes suggestive of ongoing acute or recent (<48 hours) myocardial infarction.
* Angiographic evidence of a de novo lesion > 50% requiring implantation of two DES in overlapping with a total stent length > 33 mm and reference vessel diameter between 2.5 and 4.0 mm (by visual estimation) in one coronary vessel. Multiple lesions in the same vessels can be included but at least one lesion should require implantation of two DES in overlapping with a total stent length > 33 mm. The definition of multivessel disease requires an intention to treat at least two lesions (with a least one with the characteristics reported above) in two different major epicardial segments. For example, the presence of a lesion in the left anterior descending artery and in the obtuse marginal or the presence of a lesions in the right postero-lateral branch and in a diagonal branch will qualify as multivessel. The presence of lesions in the left anterior descending artery and in the diagonal branch will not qualify as multivessel. Bifurcation lesions and ostial lesions can be included, but only if at least two DES in overlapping with a total stent length > 33 mm are implanted in the same branch. When treating diffuse lesion in the same vessel, overlapping stenting is recommended with high pressure (>14 atm post-dilation) of the overlap zone. There is no maximum stent length to treat one coronary vessel.

Exclusion Criteria:

* Female sex with childbearing potential
* Age <18 years
* Ongoing or recent episode (<48 hours) of unstable coronary artery disease (including both ST-elevation and non-ST-elevation acute coronary syndromes)
* Administration of any GP IIb/IIIa inhibitors during the previous 2 weeks
* Serum creatinine >2.5 mg/dl or with a creatinine clearance <40mL/min
* Ongoing serious bleeding or bleeding diathesis
* Previous stroke in the last 6 months
* Major surgery within the previous 6 weeks
* Platelet count <100,000 per mm3
* Ejection Fraction below 30%
* The patient has a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, or sensitivity to contrast which cannot be adequately pre-medicated.
* Hemodynamic instability (systolic blood pressure < 100 mm Hg; heart rate < 40 bpm or >100 bpm; complex ventricular arrhythmias; AV block) requiring balloon counterpulsation or inotropic support.
* The patient is simultaneously participating in another device or drug study. Patient must have completed the follow-up phase of any previous study at least 30 days prior to enrolment in this study.
* Positive clinical history for intracranial neoplasia, AV malformation, aneurysm.
* INR ≥ 2.0 or prothrombin time 1.2 times upper limit of normality
* Clinically manifested reduced liver function
* Programmed surgery within six months

Angiographic Exclusion Criteria:

* DES implantation in a chronic total occlusion or for the treatment of in-stent restenosis.
* Treatment of lesions where the operator feels necessary the usage of rotactional atherectomy
* Vessel size < 2.25 mm or > 5 mm (by visual estimation).
* Previous implantation of a bare/DES in the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mediolanum Cardio Research, Milan, Italy